CLINICAL TRIAL: NCT07240194
Title: The Efficacy and Safety of Glofitamab in Combination With PD-1 Antibody and Lenalidomide in Patients With Relapsed/Refractory Large B-cell Lymphoma (LBCL) With TP53 Aberrations: A Prospective, Multicenter, Phase II Clinical Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, WEI XU, M.D, The First Affiliated Hospital with Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-SR-499
Record Dates: First submitted 2025-09-25; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Large B-cell Lymphoma; TP53
MeSH Terms: interventions — glofitamab; Immune Checkpoint Inhibitors; Lenalidomide; obinutuzumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Glofitamab + PD-1 Inhibitor + Lenalidomide (Experimental): This arm involves a single-arm experimental treatment where participants receive a combination therapy of glofitamab (administered with stepwise dose escalation), a PD-1 inhibitor, and Lenalidomide. The regimen is designed for participants with TP53-aberrant relapsed or refractory large B-cell lymphoma (R/R LBCL). Obinutuzumab may be administered on Day 1 of the first treatment cycle for pretreatment.
  Interventions: Drug: Glofitamab; Drug: PD-1 Inhibitor; Drug: Lenalidomide; Drug: Obinutuzumab

INTERVENTIONS:
Drug: Glofitamab — glofitamab is a CD20xCD3 T-cell-engaging bispecific antibody administered intravenously with stepwise dose escalation during the treatment period to reduce the risk of cytokine release syndrome (CRS).
Drug: PD-1 Inhibitor — A PD-1 immune checkpoint inhibitor given to enhance T-cell activation and immune-mediated tumor cell killing. Administered according to the study schedule.
Drug: Lenalidomide — Lenalidomide, an immunomodulatory agent, is administered orally during the treatment cycles to potentiate anti-tumor activity and possibly enhance the activity of both glofitamab and the PD-1 inhibitor.
Drug: Obinutuzumab — Obinutuzumab, an anti-CD20 monoclonal antibody, is administered intravenously on Day 1 of Cycle 1 as a pretreatment to mitigate immune activation effects and reduce the risk of CRS before starting glofitamab.

SUMMARY:
This is a Phase II, open-label, single-arm, multicenter study designed to evaluate the safety and efficacy of a novel combination therapy-Glofitamab, a PD-1 inhibitor, and Lenalidomide (Glofit-PD-1-Len)-in patients with TP53-aberrant relapsed or refractory large B-cell lymphoma (R/R LBCL). The study will enroll 24 participants and utilize a Simon two-stage design to assess the best complete response rate (BCR), defined as achieving complete remission (CR) per 2014 Lugano criteria during the treatment period. Secondary endpoints include overall response rate (ORR), progression-free survival (PFS), overall survival (OS), duration of response (DoR), and MRD negativity rate at the end of treatment. Safety and tolerability will also be evaluated. This study addresses a critical unmet need for patients with TP53-mutant R/R LBCL, who typically have a poor prognosis under current treatment options.

DETAILED DESCRIPTION:
This is a Phase II, open-label, single-arm, multicenter study designed to evaluate the safety and efficacy of the Glofitamab-PD-1 inhibitor-Lenalidomide combination therapy (Glofit-PD-1-Len) in patients with TP53-aberrant relapsed or refractory large B-cell lymphoma (R/R LBCL). The study aims to investigate whether this novel therapeutic combination can effectively address the high unmet medical need in this patient population, characterized by poor prognosis and resistance to standard treatments.

The study employs a Simon two-stage design, enrolling a total of 24 participants. In Stage I, an initial cohort of 9 patients will be treated and evaluated. If fewer than 2 patients achieve complete response (CR) per 2014 Lugano criteria (as verified by FDG-PET imaging), the study will be terminated early. If the threshold is met, an additional 15 patients will be recruited in Stage II for further evaluation, bringing the total to 24 patients. The primary endpoint is the best complete response rate (BCR) achieved during the treatment cycle. Secondary endpoints include overall response rate (ORR), progression-free survival (PFS), overall survival (OS), duration of response (DoR), duration of complete remission (DoCR), transplantation rate, and minimal residual disease (MRD)-negative rate at the end of treatment.

The treatment process consists of an induction stage following a screening period of up to 28 days. On Day 1 of the first treatment cycle, patients will receive pretreatment with Obinutuzumab, followed by Glofitamab with stepwise dose escalation, combined with the PD-1 inhibitor and Lenalidomide. Efficacy assessments will occur at predefined time points using Lugano response criteria. The safety of the Glofit-PD-1-Len regimen will be closely monitored, and adverse events will be recorded and graded per CTCAE version 5.0.

Patients will be excluded if they meet criteria such as prior organ transplant, recent exposure to other investigational treatments, or significant comorbid conditions, including active infections and uncontrolled autoimmune diseases. Concomitant therapies, such as corticosteroids (except for specific indications), experimental therapies, and live vaccines, are prohibited. Prophylactic measures for tumor lysis syndrome (TLS), nausea, vomiting, and diarrhea, as well as granulocyte colony-stimulating factor (G-CSF) support, will be implemented as per institutional guidelines.

The risk-benefit profile of this combination is supported by prior studies demonstrating the efficacy and acceptable safety of Glofitamab in combination therapies for LBCL. Given the significant treatment gap for TP53-aberrant R/R LBCL patients, this research seeks to advance outcomes through an innovative therapeutic approach.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form before any study-specific procedures.
* Age ≥ 18 years at the time of consent.
* Histologically confirmed large B-cell lymphoma (LBCL) with CD20 expression, including but not limited to:Diffuse large B-cell lymphoma not otherwise specified (DLBCL-NOS),Transformed follicular lymphoma (tFL),Grade 3B follicular lymphoma (3B FL),High-grade B-cell lymphoma (HGBCL),Intravascular large B-cell lymphoma (IVLBCL),Primary mediastinal large B-cell lymphoma (PMBCL),Epstein-Barr virus-positive LBCL (EBV+ LBCL).
* Relapsed or refractory (R/R) LBCL defined as:

Relapsed: Disease recurrence after achieving remission for longer than 6 months after completing the last line of therapy.

Refractory: Failure to achieve remission or progression within 6 months after completing the last line of therapy.

* Confirmed TP53 deletion or mutation via FISH or NGS.
* Not eligible for autologous stem cell transplantation (ASCT) per any of the following criteria: Age ≥ 70 years, End-stage organ dysfunction, ECOG performance status of ≥ 2,Patient decision to decline ASCT, Other investigator-determined comorbidities (e.g., severe heart or lung disease, active infections) per local clinical practice standards.
* Measurable disease at baseline, with at least:

One lymph node lesion ≥ 1.5 cm (in the longest diameter), or One extranodal lesion ≥ 1.0 cm (in the longest diameter).

* ECOG performance status of 0, 1, or 2.
* Life expectancy of ≥ 12 weeks, as assessed by the investigator.
* Adequate hematologic function unless due to extensive bone marrow involvement or spleen-related complications caused by lymphoma, defined as:

Absolute neutrophil count (ANC) ≥ 1.0 × 10⁹/L,Platelets ≥ 50 × 10⁹/L,Hemoglobin ≥ 80 g/L.

-Willingness to adhere to the study procedures, including contraception requirements during the trial for participants of reproductive potential.

Exclusion Criteria:

* Prior allogeneic stem cell transplantation or organ transplantation. Active central nervous system involvement by lymphoma. Active autoimmune diseases requiring immune suppressive therapy. Uncontrolled systemic infections, including active hepatitis B, hepatitis C, or HIV infection.

Previous treatment with Glofitamab, another bispecific antibody targeting CD20 and CD3, or PD-1 inhibitors combined with Lenalidomide.

History of severe hypersensitivity to monoclonal antibodies or any components of the study drugs.

Concurrent participation in another investigational study. Use of systemic immunosuppressive therapy within 14 days prior to enrollment (excluding corticosteroids for lymphoma treatment or prevention of adverse effects).

Pregnant or breastfeeding women. Any psychological, social, or medical condition that, in the investigator's opinion, could interfere with study compliance or compromise the participants' safety or outcome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Best Complete Response Rate (BCR) | Up to 18 months after the first dose
  The proportion of participants who achieve a best complete response (CR) during the treatment period, as assessed by the 2014 Lugano criteria using FDG-PET imaging.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 18 months after the first dose
  The proportion of participants who achieve an overall response (complete response or partial response) during the treatment period, as assessed by the 2014 Lugano criteria.
Progression-Free Survival (PFS) | Time from the first dose to disease progression or death, assessed up to 24 months
  The length of time during and after treatment that the participant lives without progression of the disease, as assessed by 2014 Lugano criteria.
Overall Survival (OS) | Time from the first dose to death from any cause, assessed up to 24 months
  The length of time from the start of treatment until death from any cause.
Duration of Response (DoR) | From the date response is first documented to the date of disease progression or death, up to 24 months
  The interval from the initial documentation of response (CR or PR) to the first documentation of disease progression or death.
Duration of Complete Remission (DoCR) | From the date complete response (CR) is first documented to the date of disease progression or death, up to 24 months
  The interval from the initial documentation of CR to the first documentation of disease progression or death.
Incidence of Treatment-Related Adverse Events (Safety and Tolerability) | Up to 24 months
  The incidence, type, and severity of adverse events (graded according to CTCAE v5.0), and their relationship to the study treatment.

OTHER OUTCOMES:
Minimal Residual Disease (MRD)-Negative Rate | At the end of treatment, approximately 20 months
  The proportion of patients who achieve minimal residual disease negativity at the completion of treatment.
Transplantation Rate | Up to 12 months after the first dose
  The proportion of patients who successfully undergo stem cell transplantation after achieving remission with the study treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China